CLINICAL TRIAL: NCT06436066
Title: Effect of Self-Acupressure Application on Peripheral Neuropathic Pain and HbA1c in Patients With Type 2 Diabetes
Brief Title: Effect of Self-Acupressure on Peripheral Neuropathic Pain and HbA1c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EAVSAR
Record Dates: First submitted 2024-05-14; First posted 2024-05-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Self-acupressure; HbA1c; Peripheral Neuropathic Pain
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): A self-acupressure training booklet was created in line with the relevant literature. For the training booklet, expert opinions were received from 5 clinician nurses and 5 academic nurses who are experts in their fields. The training booklet includes the definition of self-acupressure, the areas in which it is used, its benefits, the purpose of the study, the points where acupressure will be applied and the application procedure. After 30 minutes of self-acupressure training was given to the patients in the intervention group, the relevant training booklet was delivered. Reminder messages will be sent to patients every week. They will be asked to do it 3 days a week and for 3 months. They were informed to come for a check-up after 3 months.
  Interventions: Other: Self-Acupressure
- Control Group (No Intervention): Routine clinical care continued to be provided to the patients in the control group.
  Routine maintenance applications include the following parameters;
  1. Patient Information Form
  2. Neuropathic Pain Questionnaire - DN4
  3. Neuropathic Pain Questionnaire - Short Form
  4. Providing acupressure training to diabetic patients who wish to do so at the end of the study.

INTERVENTIONS:
Other: Self-Acupressure — Applications include the following parameters;
  1. Patient Information Form (before and after application)
  2. Neuropathic Pain Questionnaire - DN4 (before and after application)
  3. Neuropathic Pain Questionnaire - Short Form (before and after application)
  4. Providing self-acupressure training (before application)
  5. Delivery of the self-acupressure training booklet (before application)
  6. Sending weekly reminder messages (during implementation)
  7. Calling the patient for a check-up after 3 months and re-evaluating with the same scales (After the application)
  8. Self-Acupressure - Satisfaction Evaluation Form with Visual Analogue Scale (After application)
  Arms: Intervention Group

SUMMARY:
Aim: This study was conducted to examine the effect of self-applied acupressure on HbA1c and peripheral neuropathic pain in patients diagnosed with type 2 diabetes.

Background: Acupressure is an effective method for relieving pain, and this effectiveness is explained by the gate control theory and endorphin theory. There is only one study in the literature showing that acupressure reduces diabetic neuropathic pain. However, in this study, acupressure was performed by a trained health professional, not by the patient himself. Measurement of glycosylated hemoglobin (HbA1c) level is one of the standard methods for long-term management of diabetes and indicates the average blood glucose concentration over a three-month period. As a result of a meta-analysis study conducted in 2023, it was reported that acupressure significantly reduced the HbA1c level.

Design: This study was designed as a randomized controlled and experimental type study.

Methods: The study is conducted with patients with type 2 diabetes who are followed in the diabetes outpatient clinic of a training and research hospital between May-November 2024. There are 2 arms in the study. The study is conducted with a total of 60 patients, 30 in the control group and 30 in the intervention group. Data collection tools are "Patient Information Form", "Neuropathic Pain Questionnaire - DN4", "Neuropathic Pain Questionnaire - Short Form" and "Self-Acupressure - Satisfaction Evaluation Form with Visual Analogue Scale". While patients in the control group continue to receive routine care, patients in the intervention group are given self-acupressure training. Patients who receive training perform acupressure on their own 3 days a week for 3 months and record it on the follow-up form.

DETAILED DESCRIPTION:
Patients with diabetes need to maintain many factors such as appropriate lifestyle changes, nutrition regulation, exercise, regular use of medications and insulin in order to prevent the emergence of peripheral neuropathy and various symptoms that develop accordingly or to control the current problem. Patients with diabetes are increasingly turning to complementary medicine methods to support such a complex process. One of these methods is acupressure, which does not involve any invasive procedures. Acupressure regulates blood flow by providing vasodilation and reduces the release of epinephrine and norepinephrine. Acupressure is a safe technique because it is a non-invasive practice. There is only one study in the literature examining the effect of acupressure on diabetic peripheral neuropathic pain, but the method used in this study is not self-acupressure, but acupressure applied by a healthcare professional. There are also studies showing that acupressure reduces plasma blood glucose levels. Self-acupressure is a method that has no side effects, is simple, convenient, does not require special equipment, and can be applied cost-effectively by trained individuals. Nurses can easily learn acupressure, apply it in clinics to increase patients' comfort and reduce symptoms, and teach patients to apply it on their own. When a person learns how to apply acupressure on his own, he needs less help to complete his treatment.This study, which was conducted to determine whether self-applied acupressure by patients diagnosed with type 2 diabetes has an effect on HbA1c and peripheral neuropathic pain, will add innovation to the literature, will guide new research in this context, and can alleviate diabetic peripheral neuropathic pain thanks to self-acupressure training given to the patient. It is thought that it will provide blood glucose level regulation and sustainability, reduce the frequency of admission to healthcare institutions and be a cost-effective application.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Diagnosed with type-2 diabetes,
* Diagnosed with peripheral neuropathy,
* DN4 score ≥ 4,
* Not diagnosed with a psychiatric disease,
* No hearing, visual or physical disabilities
* Knowing how to read and write,
* Able to communicate, no language problems,
* Having the equipment (smartphone, computer, tablet, etc.) to watch self-acupressure videos and receive reminder text messages,
* Patients who volunteer to participate in the study and give verbal and written consent will be included in the study.

Exclusion Criteria:

* Presence of lesion/scar/mass/open wound at the point where acupressure will be applied,
* Having a non-diabetic disease that causes neuropathy,
* Starting to use new medication to control neuropathic symptoms,
* Changing the dose of the current drug used to control neuropathic symptoms (if it is used routinely and the dose will not be changed, it can be included in the study),
* Adding a new oral antidiabetic drug to your current treatment,
* Not using insulin normally and starting a new insulin treatment,
* The need for a new insulin dose adjustment in insulin users (individuals who currently use insulin and whose dose will not be changed can be included in the study),
* Failure to comply with planned initiatives,
* Using psychiatric medication,
* Having a visual or hearing impairment,
* Having a mental disability or perception problem,
* Already doing self-acupressure,
* Not being willing to participate in the study is a criterion that will exclude individuals from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | First day and 3th months
  The form prepared by the researcher includes questions inquiring about the sociodemographic and background information of the patients, clinical characteristics and laboratory results.
Neuropathic Pain Questionnaire - DN4 | First day and 3th months
  In the survey, neuropathic pain is evaluated with questions based on interview with the individual and clinical examination. The highest score that can be obtained is 10. The cutoff value for neuropathic pain is accepted as 4/10.
Neuropathic Pain Questionnaire - Short Form | First day and 3th months
  Tingling, numbness and pain that increases with touch are evaluated. If the obtained scores are analyzed according to the calculation instructions, the result will reveal whether the pain in the individual is neuropathic or not.
Self-Acupressure - Satisfaction Evaluation Form with Visual Analogue Scale | 3th months
  Visual Analogue Scale (VAS) will be used to evaluate patients' satisfaction with acupressure self-administration. In the scale, a score of "1" indicates that they are not satisfied with self-acupressure, a score of "5" indicates that satisfaction is at a medium level, a score of "10" indicates that satisfaction is very high, and as the score increases, it will be stated that satisfaction increases. Patients will be asked to self-rate their acupressure satisfaction level.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Çelik, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Yeditepe University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: article — https://ebcj.mums.ac.ir/http:/ebcj.mums.ac.ir/article_21893.html
- See also: article — https://pubmed.ncbi.nlm.nih.gov/30431314/
- See also: article — https://pubmed.ncbi.nlm.nih.gov/31613424/
- See also: article — https://pubmed.ncbi.nlm.nih.gov/31758688/
- See also: article — https://pubmed.ncbi.nlm.nih.gov/17641562/
- See also: article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6122868/
- See also: article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8053207/
- See also: article — https://pubmed.ncbi.nlm.nih.gov/33894577/